CLINICAL TRIAL: NCT03185663
Title: Pilot Study Comparing Two Techniques of Taking Care Analgesic in Patients 70 and Older, Awaiting Surgery After Extracapsular Fracture of the Proximal Femur
Acronym: ALGOFRACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: I15010 / ALGOFRACT
Record Dates: First submitted 2017-06-12; First posted 2017-06-14 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2020-11

CONDITIONS: Femoral Fractures
MeSH Terms: conditions — Femoral Fractures

STUDY DESIGN:
Intervention Model Description: a pillow between the legs versus traction-stuck
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- a pillow between the legs (Placebo Comparator)
  Interventions: Other: a pillow between the legs
- traction-stuck (Experimental)
  Interventions: Other: traction-stuck

INTERVENTIONS:
Other: traction-stuck — continuous pulling method: tensile force is exerted directly on the skin by means of adhesive strips, connected to weight
  Arms: traction-stuck
Other: a pillow between the legs — setting up a pillow between the legs before the care
  Arms: a pillow between the legs

SUMMARY:
The fracture of the proximal femur is a common traumatic pathology in patients aged over 70 years, associated with a mortality of 20 to 30% a year. The care is delayed emergency. During this wait, the occurrence of heel pressure ulcers is regularly found, despite wearing antiescarres slippers. Mobilization, source of pain, is also problematic.

759/5000

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 70 and over,
* Extracapsular fracture isolated from the proximal end of the femur,
* Informed consent of the patient for participation in the study,
* Patient affiliated to a social security scheme.

Exclusion Criteria:

* Restlessness or fragile skin condition that may prevent the establishment or maintenance of traction stuck preoperatively
* Insane or confounding Pathology,
* Predictable time before operation> to 72 hours (eg anticoagulated patient orally before the fracture [antiplatelet agents are allowed], other associated diseases: urinary tract infection, pneumonia ...)
* Patient under guardianship, curatorship, or under judicial protection.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2021-05-25 (Actual)

PRIMARY OUTCOMES:
Score from pain immediately after washing, the day of surgery preoperatively | 5 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Limoges Hospital, Limoges, France

IPD SHARING:
Plan to Share IPD: No